CLINICAL TRIAL: NCT06357377
Title: An Open Label, Phase 1b Safety, Dose-finding, Brain Tumor Delivery, and Pharmacokinetics Study of Intranasal NEO100 in Patients With Pediatric-type Select Brain Tumors
Brief Title: A Study of the Safety, Dosing, and Delivery of NEO100 in Patients With Pediatric Brain Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Neonc Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO100-03
Record Dates: First submitted 2024-03-13; First posted 2024-04-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Tumor of CNS; Pediatric Tumor of Brain; Diffuse Midline Glioma, H3 K27M-Mutant; Pediatric Tumor of Brain Stem; Pineocytoma; Choroid Plexus Carcinoma, Childhood; Spinal Cord Tumor; High Grade Glioma
Keywords: High grade glioma; Diffuse Midline Glioma; H3 K27-altered; Diffuse hemispheric glioma; H3 G34-mutant; Diffuse pediatric-type HGG; H3-wildtype; IDH-wildtype; spinal cord tumors; Brainstem; Posterior fossa; Choroid plexus carcinoma; CNS embryonal tumors; Pineoblastoma; NEO100
MeSH Terms: conditions — Central Nervous System Neoplasms; Pinealoma; Choroid Plexus Carcinoma; Spinal Cord Neoplasms; Glioma | interventions — perillyl alcohol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1b safety, dose finding, brain-tumor delivery, and pharmacokinetics of IN NEO100 (Experimental): Patients will receive IN NEO100 that will follow a dose titration design, followed by a standard dose escalation design to establish safety. Brain tumor delivery of NEO100 will be confirmed in each disease sub-type by surgical resection/needle biopsy only if clinically indicated and scheduled for clinical purposes and testing with residual tissue for NEO100 and the major metabolite of NEO100 (Perillic Acid).
  The study will use a modified Fibonacci dose titration design, followed by a standard dose escalation design.
  * Cohort 1: 192 mg NEO100, QID on a 28-day cycle
  * Cohort 2: 288 mg NEO100, QID on a 28-day cycle
  * Cohort 3: 384 mg NEO100, TID on a 28-day cycle;
  * Cohort 4 (ceiling dose): 576 mg NEO100, BID on a 28-day cycle.
  Patients undergoing surgical or needle biopsy (only when clinically indicated) will receive a minimum of four days IN NEO100 treatment prior to the procedure.
  Interventions: Drug: NEO100

INTERVENTIONS:
Drug: NEO100 — NEO100 is a purified form (>98.5%) of the naturally occurring monoterpene perillyl alcohol.
  NEO100 drug product is a non-sterile solution for intranasal administration. It is compounded as a 10% solution in a 50:50 mixture of ethanol:glycerol.

SUMMARY:
This is an open label, Phase 1b safety, dose-finding, brain tumor delivery, and pharmacokinetics study of intranasal NEO100 in patients with pediatric-type diffuse high grade gliomas. Patients will receive IN NEO100 that will follow a dose titration design, followed by a standard dose escalation design to establish safety. Brain tumor delivery of NEO100 will be confirmed in each disease sub-type by surgical resection/needle biopsy only if clinically indicated and scheduled for clinical purposes and testing with residual tissue for NEO100 and the major metabolite of NEO100 (Perillic Acid).

DETAILED DESCRIPTION:
NEO100 drug product is a non-sterile solution for intranasal administration.

A feature of the clinical trials of NEO100 is to investigate the efficacy of this drug when it is delivered intranasally. Based on the general body of data on intranasal drug delivery, as well as the promising results from clinical studies in which perillyl alcohol was delivered intranasally, NeOnc expects that intranasal administration of NEO100 will allow rapid and more selective delivery of therapeutic levels of the drug to the brain, while minimizing systemic toxicity and first pass metabolism.

The study is a dose titration 1+1 design with a modified Fibonacci dose escalation, followed by a expansion design, used to determine the maximum tolerated dose and to select a recommended Phase 2 dose (RP2D). The starting dose of 192 mg mg/dose administered QID, on a 28-day cycle, is one dose below the safe dose administered to adults in a Phase 1/2a study. Dosing will increase using a modified Fibonacci dose escalation. The daily dose will start at 768 mg/day, and rise to 1,152 mg/day, which is also the safe dose administered to adults in a Phase 1/2a study.

The study is open to patient with Pediatric-type high grade glioma: Newly diagnosed and recurrent Diffuse Midline Glioma, H3 K27-altered; Diffuse hemispheric glioma, H3 G34-mutant, grade III and IV diffuse pediatric-type HGG, H3-wildtype and IDH-wildtype (including spinal cord tumors); Recurrent malignant tumors involving the brainstem or posterior fossa (choroid plexus carcinoma, CNS embryonal tumors, and pineoblastoma).

ELIGIBILITY:
Inclusion Criteria:

* Patient must have radiographically confirmed, newly diagnosed or recurrent pediatric-type high grade glioma: Diffuse Midline Glioma, H3 K27-altered; Diffuse hemispheric glioma, H3 G34-mutant, Diffuse pediatric-type HGG, grade III and IV H3-wildtype and IDH-wildtype with imaging and/or pathology consistent with a DMG, (including spinal cord tumors); or Recurrent malignant tumors involving the brainstem or posterior fossa (choroid plexus carcinoma, CNS embryonal tumors, and pineoblastoma).
* Karnofsky ≥ 50 for patients > 16 years of age or Lansky ≥ 50 for patients ≤ 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* If clinically indicated, participants must be willing to provide adequate tissue for PK analysis, either from a surgical biopsy or needle biopsy.
* Aged ≥5 to ≤18 years.
* Patients recurrent or progressive disease must have recovered from all acute side effects of prior therapy.
* From the projected start of scheduled study treatment, the following time periods must have elapsed: At least 7 days after last dose of a biologic agent or beyond time during which adverse events are known to occur for a biologic agent, 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies.
* Prior use of temozolomide during radiation at maximum of the standard pediatric dosing (defined as 90 mg/m2 /dose continuously during radiation therapy for 42 days) or dexamethasone is allowed.
* Corticosteroids: Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 3 days prior to baseline magnetic resonance imaging (MRI) scan.
* Surgical Resection: Patients may not have had a surgical resection within four weeks of starting NEO100 and any post-surgical complications must have resolved prior to initiation of NEO100.
* Radiation Therapy: Patients may not receive radiation therapy within four weeks of starting NEO100. Patients may not be enrolled if they require radiation therapy during Cycle 1 (the DLT Period). Patients may have SOC radiation therapy in Cycle 2 or beyond but will require a second DLT evaluation period to participate.
* Peripheral absolute neutrophil count (ANC) ≥ 1000/mm^3 (1.0g/l) AND
* Platelet count ≥ 100,000/mm^3 (100x10^9/l) (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m^2.
* Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age.
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase (ALT)) ≤ 2 x ULN.
* Serum albumin ≥ 2 g/dL.
* No or mild renal impairment (i.e., 60 mL/min or 1.73m2 with Schwartz equation).
* No evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and a pulse oximetry of > 92% while breathing room air.
* Participants with seizure disorder may be enrolled if seizure disorder is well controlled.
* The effects of the study drugs on the developing human fetus are unknown. For this reason, females of child-bearing potential and males must agree to use adequate contraception. Adequate methods include: hormonal or barrier method of birth control; or abstinence prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Males treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of study participation.
* A legal parent/guardian and patient must be able to understand, and willing to sign, a written informed consent (parental permission) or assent document, as appropriate.

Exclusion Criteria:

* Diagnosis of any pediatric-type glioma not described in inclusion criteria.
* Participants who are currently receiving another investigational drug. Investigational imaging agents or agents used to enhance tumor visibility on imaging or during tumor biopsy/resection should be discussed with the Medical Monitors.
* Participants who are currently receiving other anti-cancer agents.
* Participants with a known disorder that affects their immune system, such as human immunodeficiency virus (HIV) or hepatitis B or C, or an auto-immune disorder requiring systemic cytotoxic or immunosuppressive therapy. Note: Participants that are currently using inhaled, intranasal, ocular, topical or other non-oral or non-intravenous (IV) steroids are not necessarily excluded from the study but need to be discussed with the Medical Monitor.
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds (ms).
* A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome), or the use of concomitant medications that prolong the QT/QTc interval.
* Participants with uncontrolled infection or other uncontrolled systemic illness.
* Female patients of childbearing potential must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test prior to the start of therapy (as clinically indicated).
* Active illicit drug use or diagnosis of alcoholism.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as the agents used in study.
* Evidence of disseminated disease, including diffuse leptomeningeal disease or evidence of CSF dissemination as determined based upon available clinical details and not a study required MRI study or CSF test.
* Known additional malignancy that is progressing or requires active treatment within 3 years of start of study drug.
* Concomitant use of potent CYP3A4/5 inhibitors during the treatment phase of the study and within 72 hours prior to starting study drug administration.
* Concomitant use of potent CYP3A4/5 inducers, which include enzyme inducing antiepileptic drugs (EIAEDs), during the treatment phase of the study and within 2 weeks prior to starting treatment. Concurrent corticosteroids are allowed.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Nature and severity of adverse events | 6 months
  Assess the safety and tolerability of increasing dose levels of intranasally administered NEO100 using the NCI CTCAE (version 5.0) for reporting of non-hematologic AEs

SECONDARY OUTCOMES:
Identify the maximum tolerated dose (MTD) of NEO100 | 6 months
  Assess the maximum tolerated dose (MTD) of intranasally administered NEO100 using the NCI CTCAE (version 5.0) for reporting of non-hematologic AEs
Determine the recommended Phase 2 dose (RP2D) of NEO100 | 6 months
  Assess the maximum tolerated dose (MTD) of intranasally administered NEO100 using the NCI CTCAE (version 5.0) for reporting of non-hematologic AEs
Measurement of NEO100 and its metabolite perillic acid in brain tumor tissue | 6 months
  Confirm brain tumor delivery by measuring levels of NEO100 (POH) and its metabolite perillic acid (PA) in postsurgical tumor tissue in patients with pediatric-type brain tumors (measured in ng/mg).
Blood brain barrier penetration | 6 months
  To confirm blood brain barrier (BBB) penetration of NEO100 by measuring the concentration of NEO100 and its metabolite in resected tumor tissue.
Characterize the pharmacokinetics (PK) of NEO100 as measured by Peak Plasma Concentration | 6 months
  Pharmacokinetic parameters of NEO100 metabolite perillic acid in the resected tumor tissue as measured by peak plasma concentration (Cmax).
Characterize the pharmacokinetics (PK) of NEO100 as measured by the Time to Peak Plasma Concentration | 6 months
  Pharmacokinetic parameters of NEO100 metabolite perillic acid in the resected tumor tissue as measured by the time to peak plasma concentration (Tmax).
Characterize the pharmacokinetics (PK) of NEO100 as measured by Area Under the Curve | 6 months
  Pharmacokinetic parameters of NEO100 metabolite perillic acid in the resected tumor tissue as measured by the area under the plasma concentration vs time curve (AUC).
To assess efficacy of NEO100 based on objective response rate (ORR). | 6 months
  Objective CNS tumor response to NEO100 as determined by RANO 2.0 criteria.
To assess efficacy of NEO100 based on progression free survival (PFS). | 6 months
  Progression free survival (PFS).
To assess efficacy of NEO100 based on overall survival (OS). | 6 months
  Overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chen, MD, PhD, Study Chair — NeOnc Technologies Holdings, Inc.; Josh Neman, PhD, Study Director — NeOnc Technologies Holdings, Inc.

IPD SHARING:
Plan to Share IPD: Undecided